CLINICAL TRIAL: NCT01607788
Title: Prospective Database of Liver Transplantation for Hepatocellular Carcinoma
Brief Title: Prospective Liver Tumor (ProLiT) Database
Acronym: ProLit
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Geneva, Switzerland (Other)
Collaborators: University of Alberta (Other); London Health Sciences Centre (Other); University of Bern (Other); University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Christian Toso, Médecin Adjoint Agrégé, University of Geneva, University of Geneva, Switzerland
Other Study IDs: ProLit
Record Dates: First submitted 2012-05-24; First posted 2012-05-30 (Estimated); Last update posted 2012-05-30 (Estimated); Status verified 2012-05

CONDITIONS: Hepatocellular Carcinoma; Evidence of Liver Transplantation
Keywords: Selection criteria; Liver transplantation; Hepatocellular carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The investigators propose a prospective, web-based database (developed within the framework of Quickbase, Intuit) which will allow an evaluation of the data for patients with a liver tumour who receive a liver transplant. Each site will continue to transplant according to their own criteria for inclusion on the waiting list. Each center will be responsible to enter a short list of data points at time of listing, transplant, and at 1 and 2 years post transplant. Data will be gathered prospectively through a web-based anaonymized database, and outcomes analyzed yearly X5 for tumour recurrence and patient survival.

DETAILED DESCRIPTION:
A previous retrospective study evaluated the UNOS database of liver transplant recipients for use of total tumor volume (TTV) and alphafetoprotein (AFP) as criteria for selection of candidates for liver transplantation. The results confirmed a prior publication demonstrating that tumors modestly beyond Milan size limitation and irrespective of tumor numbers can achieve excellent outcomes, while providing important insight into which tumors within Milan criteria remain with a high likelihood of recurrence (high AFP). The work has now been published in Hepatology.

The investigators propose a prospective evaluation of these composite criteria, using data from patients receiving a liver transplant in order to have a larger population. Centers will continue to transplant according to their own criteria for inclusion on the waiting list. Data will be gathered prospectively through a web-based database (Quickbase, Intuit) and outcomes analyzed yearly for 5 years follow-up for tumour recurrence and patient survival.

Each center will be responsible to enter a short list of data points for their patients at time of listing, time of transplant, and yearly post transplant. Data points have been kept to a minimum in the hope that this will encourage participation in this database.

The database will be set up with 3 levels of access:

1. data entry only (one at each site)
2. review site data and composite data from other sites(one at each site)
3. review all sites and aggregate (for analysis and publication) Sites will only be able to edit and review their own patient data. They will be able to view aggregate data from other sites from which all identifiers have been removed.

Data will not be used to manage patient care in any way. The data will be used only to evaluate outcomes of patients who had a liver tumour at the time of their liver transplant.

ELIGIBILITY:
Inclusion Criteria:

* patients with hepatocellular carcinoma listed for liver transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with hepatocellular carcinoma listed for liver transplantation at the participating centers
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2009-11; Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Post-transplant survival | 24 months post-transplant

CONTACTS AND LOCATIONS:
Overall Officials: Norman Kneteman, MD, PhD, Principal Investigator — University of Geneva
Locations (1):
- University of Alberta, Edmonton, Canada